CLINICAL TRIAL: NCT06723132
Title: A Retrospective Study of Prognostic Factors and Survival of Breast Cancer Patients with Brain Metastesis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Huda Abdelsamee Thabet Mohamed, resident doctor at Clinical oncology department, Assiut University
Other Study IDs: prognostic factors+survival BC
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: prognostic factors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- breast cancer: breast cancer patients with -Radiological documentation of BM by computed tomography (CT) OR magnetic resonance imaging (MRI)

SUMMARY:
The aim of the study is to to describe the pattern of BM in breast cancer patients, assess the prognostic significance of patient related-factors and to evaluate the efficacy of various treatment modalities. clinicopathological factors and prognostic factors that affect the occurrence of brain metastases and which factors affect the survival after the occurrence of brain metastases remain to be identified . This may help identify patients at high risk for brain metastases and patients with poor prognosis after brain metastases, thus providing them with some preventive or therapeutic measures.

DETAILED DESCRIPTION:
Breast cancer (BC) has become the malignancy with the highest morbidity rate in women. Despite significant advances in the diagnosis and treatment of breast cancer, metastasis is still an important factor that seriously affects patients' quality of life and prognosis. It has been reported that distant metastases have been found at the initial diagnosis of breast cancer in about 6-10% of patients The bones, lungs, liver and brain are the four most common distant metastatic sites of breast cancer Compared with bone metastases and visceral metastases, patients with brain metastases have significantly worse prognosis The median time from diagnosis of breast cancer to CNS metastasis has been reported to be 33 month The survival of these patients may be affected by factors including molecular subtypes, performance status, ressectability of BM and visceral metastasis burden. When detected, its treatment is usually difficult and unfortunately has reverse effects on life expectancy Multi-disciplinary therapy (MDT) is the first choice for the treatment of brain metastases in breast cancer MDT for breast cancer brain metastasis includes surgery, whole brain radiation therapy (WBRT), stereotactic radiosurgery (SRS), chemotherapy, endocrine therapy, targeted therapy, etc. For patients with multiple brain metastases and neurological symptoms, WBRT combined with palliative care is the preferred option In general, patients with brain metastases of 3 or less were recommended to receive surgical resection. Patients with 4 to 5 brain metastases but less 3cm in diameter can undergo SRS .

ELIGIBILITY:
Inclusion Criteria:

* -Age >18
* Histological proven breast cancer
* Radiological documentation of BM by computed tomography (CT) OR magnetic resonance imaging (MRI)
* Patients who had been followed up for at least 6 months.

Exclusion Criteria:

* -Not histologically proven Breast cancer
* Patient without full medical data
* Those with previous or concurrent diagnosis of second primary malignancy
* Patients with leptomeningeal or dural metastases without co-existent parenchymal metastatic lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients with brain metasets
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
overall survival time | baseline
  Time from brain metasets diagnosis till death.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamamoto M, Serizawa T, Higuchi Y, Sato Y, Kawagishi J, Yamanaka K, Shuto T, Akabane A, Jokura H, Yomo S, Nagano O, Aoyama H. A Multi-institutional Prospective Observational Study of Stereotactic Radiosurgery for Patients With Multiple Brain Metastases (JLGK0901 Study Update): Irradiation-related Complications and Long-term Maintenance of Mini-Mental State Examination Scores. Int J Radiat Oncol Biol Phys. 2017 Sep 1;99(1):31-40. doi: 10.1016/j.ijrobp.2017.04.037. Epub 2017 Aug 7. PMID 28816158